CLINICAL TRIAL: NCT05667389
Title: Evaluation of the Vascular and Neural Elements Located in the Symphyseal Region Before Implant Surgery: a Retrospective Study of Cone Beam Computed Tomography (CBCT) Scans of the Face Performed on Totally Edentulous Patients in the Odontology Department of the Rothschild Hospital
Brief Title: Evaluation of the Vascular and Neural Elements Located in the Symphyseal Region Before Implant Surgery
Acronym: NERVIMPLANT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP211120
Record Dates: First submitted 2022-11-21; First posted 2022-12-28 (Actual); Last update posted 2022-12-28 (Actual); Status verified 2022-12

CONDITIONS: Mouth, Edentulous
Keywords: Cone beam computed tomography imaging; Edentulous mandibule; Symphyseal area; Vascular; Nervous; Implant
MeSH Terms: conditions — Mouth, Edentulous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The placement of implants in the symphyseal region is common, especially in the treatment of totally edentulous patients. Some implant surgical procedures may however be responsible for lesions of the vascular and nervous elements in the symphyseal region. The prevention of vascular and nervous accidents during or after implant surgery is based on the identification of vascular and nervous elements.

Although the anatomy of the symphyseal region is rather well described in the literature, the data concerning totally edentulous patients remains fragmented. These suggest that tooth avulsion and bone resorption have an influence on the anatomy of the mandibular region, and of the vascular and nervous elements traveling in the anterior mandibular part. These modifications would be responsible for individual anatomical variations.

In order to test this hypothesis, the investigator wish to evaluate the anatomical characteristics of the vascular and nervous elements located in the symphyseal region, retrospectively, of a totally edentulous population for which the anatomy was documented in a three-dimensional way from 2013 to 2021 before the placement of dental implants.

DETAILED DESCRIPTION:
The placement of dental implants in the anterior mandibular region is considered a rather safe and predictable procedure because this region has a limited number of neurovascular elements, a relatively extensive vestibular and lingual cortical bone structure, and dense trabecular bone providing high primary stability and excellent implant survival. However, this anatomical region is not free of risks, some of which are associated with potentially fatal complications (cases of death following a hemorrhagic accident have for example been described). Many clinical cases thus illustrate complications of implant surgery in the symphyseal region such as nerve damage, bone fractures, infections, and bleeding during or after the placement of the dental implant.

Implant surgery can indeed generate nerve damage according to different mechanisms by nerve compression or dilaceration by direct contact of the drill and/or the implant with the nerve compression linked to peri-implant edema or compressed bone debris at the bottom of the drill site.irritation by release of inflammatory mediators from adjacent inflamed or necrotic bone or thermal injury (heating during implant drilling). Nerve injury is clinically manifested by symptoms of varying stage and severity depending on the severity of the injury caused to the nerve. Clinically, nerve damage to the sensory afferents of the NAI can generate sensory dysfunction such as paresthesia (abnormal sensitivity), hypoesthesia (decreased sensitivity), hyperesthesia (increased sensitivity), dysesthesia (unpleasant sensitivity that may result in pain ) or even anesthesia (complete loss of sensitivity) localized to the territory of innervation of the injured nerve. From the epidemiological point of view, the frequency of such complications would be estimated between 0 and 24% for transient lesions and between 0 and 11% for irreversible lesions. Two retrospective studies carried out with more than 1300 patients with iatrogenic lesions of peripheral trigeminal afferents observed that 13% presented with pain following implant surgery.Implant surgery would thus be the second cause of NAI lesions (18%), after wisdom tooth extraction .

In implantology, vascular effraction is most often observed after perforation of the lingual cortex of the symphyseal or posterior regions , the drill causing the tearing of the underlying vascular structures. A fracture of the internal cortex during implant surgical procedures thus increases the risk of bleeding. At the level of the symphyseal region, the lesion of the sublingual artery can for example be responsible for abundant bleeding or intraoperative hemorrhage, and/or hematoma of the floor of the mouth per or postoperative , with a risk of obstruction of the upper digestive airways. From a clinical point of view, it seems very complicated to be able to establish with certainty the origin of bleeding from the floor of the mouth and only endovascular angiography can determine its origin, which complicates the management of this type of complication.

Although the anatomy of the symphyseal region is rather well described in the literature, the data concerning totally edentulous patients remains fragmented. These suggest that the avulsion of the anterior teeth and the bone resorption have an influence on the anatomy of the mandibular region, and of the vascular and nervous elements traveling in the anterior mandibular part. These modifications would be responsible for individual anatomical variations which could constitute unfavorable anatomical conditions with damage to vascular and/or nervous elements during implant surgical procedures.

In order to test this hypothesis, the investigator wish to evaluate the anatomical characteristics of the vascular and nervous elements located in the symphyseal region within a completely edentulous population for which the anatomy has been documented in a three-dimensional way before the placement of dental implants. A better knowledge of the anatomy and anatomical variations affecting the edentulous symphyseal region would allow identification of patients for whom there is a proximity between the implantation sites and the vascular and nervous elements in the edentulous symphyseal zone.

From the information collected in the clinical files (clinical and imaging data) of patients who consulted the Odontology department of the Rothschild Hospital for an imaging assessment by cone-beam computed tomography before the installation of dental implant, the investigator want to perform a descriptive analysis of the characteristics of the vascular and nervous elements (location, dimensions, anatomical relationships) located in the edentulous symphyseal area (main objective) and to specify the anatomical characteristics (height and bone thickness of the edentulous symphyseal area.

The files of totally edentulous patients who consulted the Odontology department of the Rothschild Hospital, between September 2013 and March 2021, for an imaging assessment by volume cone beam computed tomography before the placement of dental implants will be selected. Within the imaging unit, about thirty patients consult on average per year for pre-implant cone beam computed tomography imaging. Over the period 2013-2021, the population studied is thus estimated at approximately 240 patients.

A good knowledge and evaluation of the vascular and nervous elements during the pre-implant assessment is a prerequisite for limiting the risks of per and post-operative complications. If the anatomy of the symphyseal area is rather well described in the literature in dentate subjects, few data remain available in totally edentulous patients for whom the avulsion of the teeth and the bone resorption could lead to anatomical modifications impacting the elements vasculo-nervous traveling in the edentulous symphyseal zone.

Our working hypothesis is that the vascular and nervous elements traveling in the symphyseal region of edentulous patients are numerous and often located near the implantation sites in the symphyseal region. The study project will make it possible to document and enrich anatomical knowledge by specifying the characteristics of the vasculo-nervous elements progressing at the level of the symphyseal zone in a series of totally edentulous patients followed in the department for a pre-treatment imaging assessment. implant. The analysis of these epidemiological, medical and anatomical data from the clinical records of patients will also make it possible to specify the anatomical relationships between the vascular-nervous elements and the planned implantation sites.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged > 18 years old, totally edentulous, that have benefited from a CBCT examination in the odontology department with a view to implantation in the symphyseal region from 2013 to 2021
* Not opposed to the use of their data

Exclusion Criteria:

* Non-French speaking person

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Totally edentulous patients that have consulted in the odontology department of Rothschild Hospital from September 2013 to March 2021 for an imaging assessment by Cone Beam Computed Tomography before implant placement.
Sampling Method: Non-Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2022-12 (Estimated); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Characteristics of the vascular and nervous elements located in the edentulous symphyseal area | Before implant placement (one day)
  Number and localisation of foramina location

SECONDARY OUTCOMES:
Characteristics of the vascular and nervous elements located in the edentulous symphyseal area : diameter | Before implant placement (one day)
  The diameter of the incisor canal
Characteristics of the vascular and nervous elements located in the edentulous symphyseal area : mesio-distal dimension | Before implant placement (one day)
  The mesio-distal dimension of the incisal canal
Characteristics of the vascular and nervous elements located in the edentulous symphyseal area : diameter of the opening | Before implant placement (one day)
  The diameter of the opening of the lingual foramen from the end of the lingual canal
Characteristics of the vascular and nervous elements located in the edentulous symphyseal area : vestibular and lingual position | Before implant placement (one day)
  The vestibular and lingual position of the tongue canal
Anatomical characteristics of the edentulous symphyseal area. | Before implant placement (one day)
  Height and bone thickness within the symphyseal mandibule

CONTACTS AND LOCATIONS:
Overall Officials: Adeline BRAUD, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hospital Rotschild, Odontology Department, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided